CLINICAL TRIAL: NCT01083823
Title: Calling for Care: Cell Phones for Mood Telemetry
Brief Title: Calling for Care: Cell Phones for Mood Telemetry in Teens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Motorola Canada Limited (Industry)
Responsible Party: Principal Investigator, Dr. David Kreindler, Active Staff, Sunnybrook Health Sciences Centre
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 364-2007
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Bipolar Disorder; Cyclothymia; Borderline Personality Disorder
Keywords: Mental health telemetry; Mood telemetry; Mood; Bipolar disorder; Affective instability; Cyclothymia; Electronic diaries; Mood diaries; Mood swings
MeSH Terms: conditions — Bipolar Disorder; Cyclothymic Disorder; Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-reported mood swings (Active Comparator): Participants who self-identify as experiencing severe mood swings that interfere with life.
  Interventions: Other: Mental health telemetry (MHT)
- Healthy (Active Comparator): Participants who self-identify as not experiencing mood swings in the past or at present and who deny past / present problems with substance use.
  Interventions: Other: Mental health telemetry (MHT)

INTERVENTIONS:
Other: Mental health telemetry (MHT) — Use a cell phone equipped with MHT software to complete a self-report mood symptom questionnaire daily at a fixed time of day, as well as additional discretionary questionnaires following any significantly stressful events.
  Other Names: Mood telemetry

SUMMARY:
We will modify our existing VMQ/VADIS mood telemetry software to run on a Motorola platform, and enhance it to collect information on both mood symptoms (currently covered by the VMQ/VADIS) as well as daily life stressors (currently outside the VMQ/VADIS' scope). By doing so, we will be able us to examine the role of daily stressors in the lives of teens with and without mood swings, to identify how changes in mood triggered by stressful events are similar to or different from mood changes linked to the bipolar disorder, borderline personality disorder, or other forms of affective instability.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-20yrs,
* Either (i) self-reported healthy with no past / present history of substance use problems OR (ii) self-reported severe mood swings interfering with daily life.
* Fluent in English.

Exclusion Criteria:

* Inability to be trained successfully on the MHT software or to complete questionnaires without assistance.
* Unwillingness to sign / maintain a contract with a cell phone service provider.
* Lack of parental assent / willingness to act as guarantor for cell phone provider contract

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2010-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
usability | After nine months' enrollment
  Assessment of participant drop-out and reporting rates

SECONDARY OUTCOMES:
Validity | Every three months x 9 months
  Validate that the data reported by telemetry is valid, by comparing cell phone questionnaire responses with results of standardized clinical ratings collected every-three-month via face-to-face meetings
Qualitative feedback | After nine months' enrollment
  Collect human factors engineering feedback from our participants for subsequent development work, by questioning participants at the exit interview about their experience with the cell phone and software

CONTACTS AND LOCATIONS:
Overall Officials: David M Kreindler, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada